CLINICAL TRIAL: NCT06000189
Title: The Effect of Phototherapy on Demodex Density: A Case-Control Study
Brief Title: Phototherapy: Not a Cause of Demodicosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Hasan Aksoy, Medical Doctor, Istanbul Medeniyet University
Other Study IDs: 2022/0340
Record Dates: First submitted 2023-07-28; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Demodicidosis
Keywords: Demodex, phototherapy, NBUVB, demodicosis, immunsupression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who received phototherapy for various dermatological indications: A case-control study will be conducted participants who received narrow-band ultraviolet B (NBUVB) or ultraviolet A-1 (UVA-1) therapy for various dermatological indications. Standardized skin surface biopsies (SSSB) were performed before and after phototherapy to assess Demodex density. Demographic data, medical information, and the presence of demodex-related skin conditions were recorded using a standardized form. Statistical analysis will be performed to compare the demodex densities and prevalence of demodicosis between baseline and 20th session of phototherapy.
  Interventions: Procedure: Standardized skin surface biopsies (SSSB)

INTERVENTIONS:
Procedure: Standardized skin surface biopsies (SSSB) — Skin samples will be obtained from four regions of the participants' faces, including the forehead, right cheek, left cheek, and the nose, before phototherapy and after 20 sessions of phototherapy. The SSSB will be performed as follows: a 1 cm² square will be drawn on a glass slide using a ruler. The skin areas to be sampled will be gently swabbed with a dry gauze to induce irritation by this way to obtain more mites. Then, one drop of cyanoacrylate adhesive will be dropped onto the marked area on the glass slide, and the adhesive surface of the slide will be pressed onto the skin surface for approximately one minute. Afterwards, the slide will be gently lifted, and the sampled area will be examined under a light microscope at x10 and x40 magnifications after applying immersion oil. The presence of more than five Demodex mites per square centimeter will be defined as increased Demodex density.

SUMMARY:
The purpose of this study is to determine whether there is an increase in the frequency of demodicosis and the density of Demodex mites after 20 sessions of phototherapy.

The main question(s)it aims to answer are;

* Are Demodex mites higher in patients treated with phototherapy?
* In which localization and with what intensity was demodicosis most common? Participants will be assessed using standardized skin surface biopsy technique in four localization on their face.

Researchers will compare demodex intensity per cm² to see if the phototherapy effects demodex intensity on patients.

DETAILED DESCRIPTION:
This study employee as a case-control study to compare the Demodex densities before and after 20 sessions of narrow-band ultraviolet B (NBUVB) or ultraviolet A-1 (UVA-1) therapy in patients who will receive phototherapy for any dermatological indication. The study is going to be conducted at Istanbul Medeniyet University Department of Dermatology between June 2023 and August 2023. Ethical approval was obtained from Istanbul Medeniyet University Local Ethics Committee (decision number: 2022/0340).

Demographic and medical information, including age, gender, smoking and alcohol habits, dermatological indication of phototherapy, presence of facial involvement of the relevant disease, and use of medications or cosmetic products on the face in the last week, will be obtained through a standardized form. Patients will be evaluated by the researcher for the presence of clinical conditions associated with primary/secondary demodicosis, such as acne, rosacea, perioral dermatitis, seborrheic dermatitis, folliculitis, blepharitis, or pityriasis folliculorum.

The standardized skin surface biopsy (SSSB) technique is going to be utilized to assess Demodex density. Skin samples will be obtained from four regions of the participants' faces, including the forehead, right cheek, left cheek, and the nose, before phototherapy and after 20 sessions of phototherapy. The SSSB will be performed as follows: a 1 cm² square will be drawn on a glass slide using a ruler. The skin areas to be sampled will be gently swabbed with a dry gauze to induce irritation by this way to obtain more mites. Then, one drop of cyanoacrylate adhesive will be dropped onto the marked area on the glass slide, and the adhesive surface of the slide will be pressed onto the skin surface for approximately one minute. Afterwards, the slide will be gently lifted, and the sampled area will be examined under a light microscope at x10 and x40 magnifications after applying immersion oil. The presence of more than five Demodex mites per square centimeter will be defined as increased Demodex density.

Statistical analysis will be performed using IBM Statistical Package for the Social Sciences [SPSS] v.17. Means, standard deviations, or frequencies will be calculated for relevant variables as required. Paired samples t-test will be used to compare Demodex densities, and the McNemar test will be used to compare the presence of demodicosis between pre- and post-treatment. A p-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received phototherapy for various dermatological indications

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants aged between 18 and 65 which are received narrow-band ultraviolet B (NBUVB) or ultraviolet A-1 (UVA-1) therapy for various dermatological indications
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Phototherapy: Not a Cause of Demodicosis | 4 months
  A standardized form is going to be used to collect demographic information, and details regarding smoking and alcohol habits. Additional information regarding their treatment regimens will be recorded. Furthermore patients will be evaluated for the presence of acne, rosacea, perioral dermatitis, seborrheic dermatitis, folliculitis, blepharitis, or pityriasis folicullorum, as these conditions have been associated with an increased demodicosis. After that the standardized skin surface biopsy (SSSB) technique will be performed before and after phototherapy to assess Demodex density.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Aslan Kayıran, Ass.Prof, Study Chair — Istanbul Medeniyet University; sümeyye Altıntaş Kakşi, Specialist, Study Chair — Istanbul Medeniyet University; Vefa Aslı Erdemir, Prof, Study Chair — Istanbul Medeniyet University; Yeşim Dede, Resident, Study Chair — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Turkmen D, Turkoglu G. Demodex Infestation in Patients with Rosacea. Turkiye Parazitol Derg. 2019 Dec 23;43(4):194-197. doi: 10.4274/tpd.galenos.2019.6456. PMID 31865655
- [Result] Kulac M, Ciftci IH, Karaca S, Cetinkaya Z. Clinical importance of Demodex folliculorum in patients receiving phototherapy. Int J Dermatol. 2008 Jan;47(1):72-7. doi: 10.1111/j.1365-4632.2007.03336.x. PMID 18173609
- [Result] Forton F, Seys B. Density of Demodex folliculorum in rosacea: a case-control study using standardized skin-surface biopsy. Br J Dermatol. 1993 Jun;128(6):650-9. doi: 10.1111/j.1365-2133.1993.tb00261.x. PMID 8338749
- [Result] Aytekin S. Outbreak of demodex folliculitis on the face and upper trunk during 311-nm UVB therapy for psoriasis. J Eur Acad Dermatol Venereol. 2004 Mar;18(2):236-8. doi: 10.1111/j.1468-3083.2004.00898.x. No abstract available. PMID 15009323